CLINICAL TRIAL: NCT02184338
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BIRB 1017 BS (5, 25, 100, 250, 500, and 800 mg) as a Solution in PEG 400 / 26% Ethanol Administered to Healthy Male Subjects. Placebo Controlled and Blinded at Each Dose Level
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BIRB 1017 BS as a Solution in PEG 400 / 26% Ethanol Administered to Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1187.1
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BIRB 1017 BS in single rising doses (Experimental)
  Interventions: Drug: BIBR 1017 BS powder
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBR 1017 BS powder
  Arms: BIRB 1017 BS in single rising doses
Drug: Placebo — PEG 400
  Arms: Placebo

SUMMARY:
Study to assess safety, tolerability and pharmacokinetics of BIRB 1017 BS in single rising oral doses of 5 to 800 mg in a polyethylene glycol 400 (PEG 400) / 26% ethanol solution in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 18 and <= 50 years
* BMI >18.5 and <29.9 kg/m2 (Body Mass Index)

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, haematological, oncological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (< 10 days prior to study drug administration or expected during the trial)
* Participation in another trial with an investigational drug (< 2 months prior to administration or expected during trial)
* Smoker (> 10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation or loss > 400 mL, < 1 month prior to administration or expected during the trial
* Excessive physical activities (within 5 days prior to administration or during the trial)
* Clinically relevant laboratory abnormalities
* Any electrocardiogram value outside of the reference range and of clinical relevance including, but not limited to QRS interval > 110 ms or QTcB > 450 ms or QT >500 ms
* Known hypersensitivity to the drug or its excipients
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2004-08; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability by the investigator on a 4-point scale | at day 5-10
Number of patients with adverse events | up to 25 days
Number of patients with clinically significant changes in vital signs (pulse rate, systolic and diastolic blood pressure) | up to day 10
Number of patients with abnormal changes in clinical laboratory tests | up to day 10
Number of patients with clinically relevant effect on electrocardiogram parameters | up to day 10

SECONDARY OUTCOMES:
Maximum concentration of BIRB 1017 BS in plasma (Cmax) | pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 15:00, 24:00, 34:00, and 48:00 hours after administration of study drug
Time from dosing to maximum concentration (tmax) | pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 15:00, 24:00, 34:00, and 48:00 hours after administration of study drug
Area under the concentration-time curve of the analyte in plasma ofer the time interval from 0 to the last quantifiable analyte plasma concentration (AUC0-infinity) | pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 15:00, 24:00, 34:00, and 48:00 hours after administration of study drug
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable analyte plasma concentration (AUC0-tz) | pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 15:00, 24:00, 34:00, and 48:00 hours after administration of study drug
Terminal elimination rate constant in plasma (λz) | pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 15:00, 24:00, 34:00, and 48:00 hours after administration of study drug
Terminal half-life of the analyte in plasma (t1/2) | pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 15:00, 24:00, 34:00, and 48:00 hours after administration of study drug
Mean residence time of the analyte in the body (MRT) | pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 15:00, 24:00, 34:00, and 48:00 hours after administration of study drug
Apparent oral clearance of the analyte in the plasma after oral administration (CL/F) | pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 15:00, 24:00, 34:00, and 48:00 hours after administration of study drug
Apparent volume of distribution during the terminal phase λz following an oral dose (Vz/F) | pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 15:00, 24:00, 34:00, and 48:00 hours after administration of study drug